CLINICAL TRIAL: NCT02868554
Title: Orthodontic Tooth Movement With Accelerated Invisalign Therapy Using Acceledent Aura: A Randomized Clinical Trial
Brief Title: Accelerated Invisalign Therapy in Conjunction With Acceledent Aura
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: OrthoAccel Technologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16-0167
Record Dates: First submitted 2016-08-10; First posted 2016-08-16 (Estimated); Results first posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Malocclusion
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard Invisalign Therapy (No Intervention): Patients receiving standard Invisalign therapy will be instructed to wear each aligner 24 hours day. Patients will be permitted to progress to the subsequent aligner after 14 days of compliant aligner wear.
- Accelerated Invisalign (Experimental): Patients receiving accelerated Invisalign therapy will be instructed to wear each aligner 24 hours day. Patients will be permitted to progress to the subsequent aligner after 4 days of compliant aligner wear.
  Interventions: Device: Accelerated Invisalign therapy
- Accelerated Invisalign and Vibration (Experimental): In addition to the accelerated Invisalign protocol described in Arm #2, patients will undergo intraoral vibration therapy using an AcceleDent Aura device for a duration of 20 minutes per day.
  Interventions: Device: AcceleDent Aura; Device: Accelerated Invisalign therapy

INTERVENTIONS:
Device: AcceleDent Aura — Patients receiving vibration therapy will be instructed to bite down on the AcceleDent mouthpiece, which vibrates at a .25 Newtons (25 grams) force level with a 30 Hertz frequency for 20 minutes per day.
  Arms: Accelerated Invisalign and Vibration
Device: Accelerated Invisalign therapy — Patients receiving accelerated Invisalign therapy will be instructed to wear each aligner 24 hours day. Patients will be permitted to progress to the subsequent aligner after 4 days of compliant aligner wear.
  Arms: Accelerated Invisalign; Accelerated Invisalign and Vibration

SUMMARY:
Purpose:

The objective of this study is to investigate the effects of accelerated Invisalign and vibration therapy on rate of orthodontic tooth movement, activation of inflammation biomarkers as well as pain levels experienced by orthodontic patients during the initial 12 weeks of alignment.

Participants:

Up to 30 orthodontic patients of the University of North Carolina Orthodontic Residency Program will be recruited for this study. Patients older than 18 years old will be otherwise healthy subjects previously diagnosed with malocclusion.

Procedures (methods):

Each patient will be randomly allocated into either a control group or one of two intervention groups. Patients within the control group will receive standard Invisalign therapy without vibration. Patients within the intervention groups will receive accelerated Invisalign therapy with or without vibration. Patients receiving vibration therapy will utilize an AcceleDent Aura device which provides a light vibration at .25 Newtons (N) and 30 Hertz (Hz) frequency for twenty minutes daily. Three dimensional images of each subject's dentition will be recorded five times at 0 days, 4 days, 2 weeks, 6 weeks, and 12 weeks progress visits.

DETAILED DESCRIPTION:
Align Technology©, Inc. developed Invisalign® in 1997 to meet the esthetic demands of orthodontic patients and providers. Invisalign patients receive a series of computer-assisted designed stereolithic clear retainers to incrementally resolve their malocclusion. Invisalign® and other advances in orthodontic technology such as clear aligners, ceramic brackets and lingual braces offer options to address the esthetic demands of most orthodontic patients but duration of treatment continues to be one of the most challenging aspects of practice.

In 2008, OrthoAccel Technologies©, Inc. developed the AcceleDent device to accelerate tooth movement and reduce orthodontic treatment time. Patients receiving vibration therapy are instructed to bite down on the AcceleDent mouthpiece, which vibrates at a .25 N (25 grams) force level with a 30 Hz frequency for 20 minutes per day. The theory underlying AcceleDent and the use of vibration to expedite orthodontic tooth movement started in 1892 with the studies of Julius Wolff, who discovered bone adapts to pressure loads. In 2001, Astronauts in space attempted to use the principles of Wolff's Law to maintain normal bone quality by working out and performing daily tasks while standing on a vibrating plate with the aid of elastic straps. In 2004, the effect of vibration therapy on bone density was further supported when increased bone density and strength was noted in post-menopausal women who received whole body vibration therapy. OrthoAccel claims vibration therapy using the AcceleDent device can reduce treatment time up to 50 percent by accelerating the process of bone remodeling required for orthodontic tooth movement. In 2013, despite relatively little scientific evidence, the US Food and Drug Administration (FDA) approved AcceleDent as a class II medical device and orthodontic accessory to facilitate accelerated tooth movement.

Invisalign therapy in conjunction with AcceleDent has been aggressively marketed towards the esthetically sensitive patient who, not so coincidentally, is the most concerned with duration of treatment. Some orthodontic providers using vibration therapy have deviated from the standard 2-week aligner schedule and recommend a 4-day aligner schedule. Orthodontic patients receiving accelerated Invisalign therapy in conjunction with AcceleDent claim reduced treatment time by as much as 50 percent. What is responsible for the positive results? The accelerated tooth movement might simply be the result of the accelerated Invisalign therapy, which would raise the question of whether vibration therapy and the cost associated with AcceleDent is justified. The purpose and primary specific aim of our study will be to determine the cause of the accelerated tooth movement. Because the vibration therapy is used in conjunction with an accelerated Invisalign aligner schedule, there is an assumption that the vibration therapy is promoting faster tooth movement. However, the current literature, from clinical trials, supporting the efficacy of vibration therapy on accelerated tooth movement is lacking.

Accelerated orthodontic tooth movement may offer many benefits to both, the patient and the orthodontist. Reduced treatment time reduces the burden of orthodontic treatment by decreasing risk for undesired treatment sequelae (e.g., white spot lesion, caries, gingivitis, etc) and potentially reduces the discomfort commonly associated with orthodontic treatment. Orthodontists benefit from accelerated tooth movement for multiple reasons pertaining to practice management and increased profitability. Orthodontists using accelerated treatment techniques have reported increased profit margins due to reduced chair time and increased organic growth due to differentiation of the practice.

There are also potential negative outcomes associated with accelerated orthodontic tooth movement. For the patient, there is a potential increased risk for root resorption, increased treatment fees and pain associated with treatment. At this time, there is no published data regarding the potential for orthodontic relapse following the accelerated orthodontic tooth movement. There are several publications supporting the fact that relapse is a known risk for conventional orthodontic treatment. The investigators can make the safe assumption that accelerated orthodontic treatment would be no different than conventional orthodontic therapy with regard to relapse potential. All orthodontic patients must be compliant with regard to orthodontic retention or relapse will be expected. Most orthodontists are charging between $700-800 for AcceleDent therapy in addition to the normal orthodontic fee. Finally, there is no published data regarding pain associated with accelerated Invisalign treatment.

Further, the mechanism underlying any increased orthodontic tooth movement due to vibration remains unclear. Studies on a cellular level have shown a promising but complicated mechanism of how vibration may enhance activation of various cell proliferation and differentiation molecules within the periodontal ligament (PDL) stem cells as well as increase levels of gingival inflammation biomarkers. For example, vibration therapy might accelerate breakdown of the cellular cytoskeleton, increase actinG trafficking into the nucleus, increase Runx2 gene expression, and thus facilitate bone formation. Whether this mechanotransduction mechanism can be translated into clinical tooth movement is unknown and its clinical evidence remains to be elucidated.

In this study, the investigators propose a randomized prospective clinical design to investigate effects of AcceleDent vibration therapy on the efficiency of tooth movement, on the activation of gingival crevicular fluid biomarkers and on patient discomfort in conjunction with accelerated Invisalign therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females over the age of 18 years old desiring orthodontic treatment.
2. Adult dentition with all upper and lower front teeth present and any premolar and molar combination in the upper posterior of two teeth on each side.
3. Normal pulp vitality and healthy periodontal tissues as determined by intraoral exam.
4. Good health as determined by medical history.
5. Willingness and ability to comply with study procedures, attend study visits, and complete the study.
6. The ability to understand and sign a written informed consent form, which must be signed prior to initiation of study procedures.

Exclusion Criteria:

1. Patient under the age of 18 years old
2. Women may not be pregnant. Negative urine pregnancy tests prior to exposure to cone beam imaging is required to verify pregnancy status.
3. Patients diagnosed with systemic diseases such as diabetes, hypertension (high blood pressure), temporomandibular disorders (jaw disorders), or craniofacial syndromes.
4. Severe malocclusions that would require adjunctive procedures other than Invisalign. These include impacted teeth, closure of extractions spaces.
5. Significant periodontal disease (> 4mm pocket depth or >2 mm of recession on upper anterior teeth).
6. Active caries not under care of either a dentist or periodontist.
7. Chronic daily use of any non-steroidal anti-inflammatory medication, estrogen, calcitonin, or corticosteroids.
8. History of use or current use of any bisphosphonate medication or other medication for treatment of osteoporosis.
9. Current smoker (must not have smoked in the last 6 months).
10. Failing to comply with research protocols

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-08; Primary Completion 2019-04-26 (Actual); Study Completion 2019-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ching C Ko, DDS, PhD, Principal Investigator — UNC Department of Orthodontics
Locations (1):
- UNC Department of Orthodontics, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sen B, Xie Z, Uzer G, Thompson WR, Styner M, Wu X, Rubin J. Intranuclear Actin Regulates Osteogenesis. Stem Cells. 2015 Oct;33(10):3065-76. doi: 10.1002/stem.2090. PMID 26140478
- [Background] Uribe F, Padala S, Allareddy V, Nanda R. Patients', parents', and orthodontists' perceptions of the need for and costs of additional procedures to reduce treatment time. Am J Orthod Dentofacial Orthop. 2014 Apr;145(4 Suppl):S65-73. doi: 10.1016/j.ajodo.2013.12.015. PMID 24680026
- [Background] Ojima K, Dan C, Nishiyama R, Ohtsuka S, Schupp W. Accelerated extraction treatment with Invisalign. J Clin Orthod. 2014 Aug;48(8):487-99. No abstract available. PMID 25226041
- [Background] Bowman SJ. The effect of vibration on the rate of leveling and alignment. J Clin Orthod. 2014 Nov;48(11):678-88. No abstract available. PMID 25707947
- [Background] Orr MF, Ruckart PZ. Surveillance of hazardous substances releases due to system interruptions, 2002. J Hazard Mater. 2007 Apr 11;142(3):754-9. doi: 10.1016/j.jhazmat.2006.06.121. Epub 2006 Jul 3. PMID 16920261
- [Background] Nishimura M, Chiba M, Ohashi T, Sato M, Shimizu Y, Igarashi K, Mitani H. Periodontal tissue activation by vibration: intermittent stimulation by resonance vibration accelerates experimental tooth movement in rats. Am J Orthod Dentofacial Orthop. 2008 Apr;133(4):572-83. doi: 10.1016/j.ajodo.2006.01.046. PMID 18405822
- [Background] d'Apuzzo F, Cappabianca S, Ciavarella D, Monsurro A, Silvestrini-Biavati A, Perillo L. Biomarkers of periodontal tissue remodeling during orthodontic tooth movement in mice and men: overview and clinical relevance. ScientificWorldJournal. 2013 Apr 23;2013:105873. doi: 10.1155/2013/105873. Print 2013. PMID 23737704
- [Background] Meikle MC. The tissue, cellular, and molecular regulation of orthodontic tooth movement: 100 years after Carl Sandstedt. Eur J Orthod. 2006 Jun;28(3):221-40. doi: 10.1093/ejo/cjl001. Epub 2006 May 10. PMID 16687469
- [Background] Marie SS, Powers M, Sheridan JJ. Vibratory stimulation as a method of reducing pain after orthodontic appliance adjustment. J Clin Orthod. 2003 Apr;37(4):205-8; quiz 203-4. No abstract available. PMID 12747073
- [Background] Xiong J, O'Brien CA. Osteocyte RANKL: new insights into the control of bone remodeling. J Bone Miner Res. 2012 Mar;27(3):499-505. doi: 10.1002/jbmr.1547. PMID 22354849
- [Background] Leethanakul C, Suamphan S, Jitpukdeebodintra S, Thongudomporn U, Charoemratrote C. Vibratory stimulation increases interleukin-1 beta secretion during orthodontic tooth movement. Angle Orthod. 2016 Jan;86(1):74-80. doi: 10.2319/111914-830.1. Epub 2015 Mar 26. PMID 25811245
- [Background] Nimeri G, Kau CH, Abou-Kheir NS, Corona R. Acceleration of tooth movement during orthodontic treatment--a frontier in orthodontics. Prog Orthod. 2013 Oct 29;14:42. doi: 10.1186/2196-1042-14-42. PMID 24326040
- See also: OrthoAccel Technologies growth projections — http://www.prnewswire.com/news-releases/orthoaccel-technologies-continues-trajectory-of-accelerated-growth-with-over-2500-practice-locations-300088573.html
- See also: Sample study for inflammation Biomarkers — http://www.angle.org/doi/full/10.2319/111914-830.1

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Invisalign Therapy | Accelerated Invisalign | Accelerated Invisalign and Vibration
Started | 10 | 12 | 12
Completed | 7 | 12 | 11
Not Completed | 3 | 0 | 1
Not completed — Lost to Follow-up | 3 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Data are missing for 1 participant.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Invisalign Therapy | Accelerated Invisalign | Accelerated Invisalign and Vibration | Total
Number analyzed (Participants) | 10 | 12 | 11 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.9 (13.5) | 31.3 (9.1) | 31.1 (8.5) | 32.9 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 9 | 7 | 21
  Male | 5 | 3 | 4 | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 12 | 11 | 33

OUTCOME MEASURES:

1. Primary Outcome: Little's Irregularity Index (LI) at Baseline
Description: Little's Irregularity Index is the sum of contact displacement in mm between the anterior teeth from mesial of one canine to the mesial of the contralateral canine.
Time Frame: Baseline (Week 0)
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Standard Invisalign Therapy | Accelerated Invisalign | Accelerated Invisalign and Vibration
Number analyzed (Participants) | 7 | 12 | 11
mm | 6.11 (1.24) | 6.31 (2.71) | 6.89 (2.24)

2. Primary Outcome: Little's Irregularity Index at Final Stage
Description: as for outcome 1
Time Frame: End of Study (a total of approximately 12 weeks)
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Standard Invisalign Therapy | Accelerated Invisalign | Accelerated Invisalign and Vibration
Number analyzed (Participants) | 7 | 12 | 11
mm | 4.97 (1.21) | 3.07 (2.59) | 4.52 (1.61)

3. Primary Outcome: Rate of Orthodontic Tooth Movement [Difference in Little's Irregularity Index, mm/Day]
Description: The rate of orthodontic tooth movement (Little's Irregularity Index mm/day) will be evaluated. Little's Irregularity Index is the sum of contact displacement in mm between the anterior teeth from mesial of one canine to the mesial of the contralateral canine.
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: mm/day
Arm/Group | Standard Invisalign Therapy | Accelerated Invisalign | Accelerated Invisalign and Vibration
Number analyzed (Participants) | 7 | 12 | 11
mm/day | 0.0136 (0.0057) | 0.0202 (0.0135) | 0.0243 (0.0163)
Statistical Analysis 1: Comparison: Standard Invisalign Therapy vs Accelerated Invisalign vs Accelerated Invisalign and Vibration; Test type: Superiority; p = 0.07, ANOVA; Mean Difference (Final Values) = 0.05

4. Primary Outcome: Rate of Orthodontic Tooth Movement [Total % Change of Little's Irregularity Index]
Description: The percent change in the irregularity index between the baseline and the final will be evaluated. Little's Irregularity Index is the sum of contact displacement in mm between the anterior teeth from mesial of one canine to the mesial of the contralateral canine.
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: percent change in LI
Arm/Group | Standard Invisalign Therapy | Accelerated Invisalign | Accelerated Invisalign and Vibration
Number analyzed (Participants) | 7 | 12 | 11
percent change in LI | 18.90 (7.65) | 23.71 (11.02) | 29.12 (10.77)
Statistical Analysis 1: Comparison: Standard Invisalign Therapy vs Accelerated Invisalign vs Accelerated Invisalign and Vibration; Test type: Superiority; p = 0.02, ANOVA; Mean Difference (Final Values) = 0.05

5. Secondary Outcome: Activity of Bone Turnover Markers (BTMs) During Orthodontic Tooth Movement [Quantitative Polymerase Chain Reaction (qPCR), Cycle Threshold Values (Ct)]
Description: Gingival crevicular fluid will be sampled to determine if vibratory stimulation during orthodontic tooth movement increases the activity of the Receptor Activator of Nuclear Factor-KappaB (RANK), Receptor Activator of Nuclear Factor-KappaB Ligand (RANKL) and Osteoprotegerin (OPG) cell signaling pathway.
Time Frame: 12 weeks
Population: Due to loss of key study personnel these data were not collected
Arm/Group | Standard Invisalign Therapy | Accelerated Invisalign | Accelerated Invisalign and Vibration
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Mean Patient Discomfort Score
Description: Research subjects asked to complete questionaire at Week 12 in order to determine what effect vibratory stimulation has on discomfort during orthodontic treatment. The FACES Pain Visual Analog Pain Scale was used to assess pain. Pain was assessed on a 0 (no pain) to 10 (worst pain) grading scale. Lower scores reflect lower pain levels.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Invisalign Therapy | Accelerated Invisalign | Accelerated Invisalign and Vibration
Number analyzed (Participants) | 7 | 12 | 11
score on a scale | 0.643 (0.945) | 1.583 (1.379) | 0.682 (1.230)

ADVERSE EVENTS:
Time Frame: Baseline through end of study (an approximate total of up to 12 weeks).
Arm/Group | Standard Invisalign Therapy | Accelerated Invisalign | Accelerated Invisalign and Vibration
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/10 | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-01): https://cdn.clinicaltrials.gov/large-docs/54/NCT02868554/Prot_SAP_000.pdf